CLINICAL TRIAL: NCT04390178
Title: Plasma From Individuals Who Have Recovered From Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection as Treatment for Acute COVID-19 Disease
Brief Title: Convalescent Plasma as Treatment for Acute Coronavirus Disease (COVID-19)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joakim Dillner (Other)
Collaborators: Danderyd Hospital (Other); Karolinska Institutet (Other); Karolinska University Hospital (Other)
Responsible Party: Sponsor-Investigator, Joakim Dillner, Professor of Infectious Disease Epidemiology; Director of R&D, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP1
Record Dates: First submitted 2020-04-10; First posted 2020-05-15 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
Keywords: COVID-19 convalescent plasma treatment; SARS-CoV-2 infection; Safety; Effectiveness
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Intervention Model Description: An open, non-randomised controlled, clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Convalescent plasma treatment (Experimental): All participants will receive a bag of convalescent plasma. The bag volume will be 180-200 ml. The first 10 patients will receive 1, 5, 10, 50 and 134 ml of plasma at 30 minute intervals while being closely monitored for adverse events, especially allergic reactions. The remaining twenty patients will receive the convalescent plasma as a slow infusion according to normal routines.
  Interventions: Biological: SARS-CoV-2 convalescent plasma

INTERVENTIONS:
Biological: SARS-CoV-2 convalescent plasma — Treatment with convalescent plasma (180-200ml) from individuals who have recovered from SARS-CoV-2 infection

SUMMARY:
There is currently no effective treatment for COVID-19 except best supportive care. The aim is assess the safety, tolerability and efficacy of convalescent plasma for treatment of patients with varying degrees of COVID-19 illness.

DETAILED DESCRIPTION:
Convalescent plasma has been shown to be safe and effective for treatment of several diseases. Preliminary data indicates that it is safe and effective for treatment of COVID-19. However, data is limited to small studies and case series on severely ill patients. The proposed study assesses the safety and efficacy earlier in the course of illness, in slightly less severe patients with the possibility of detecting less severe adverse events and the potential for early treatment to hinder the development of severe disease. Plasma is collected from consenting donors who have recovered from SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and <81 years
* Active COVID-19 defined as symptoms + SARS CoV-2 identified from upper or lower airway samples
* Fever ≥38.5C, admitted to a study hospital, hypoxemia defined as having a peripheral oxygen saturation below 93% (measured by pulse oximetry) and a breathing rate of >20 breaths per minute without supplemental oxygen treatment
* A negative pregnancy test taken before inclusion and use of an acceptable effective method of contraception until treatment discontinuation if the participant is a woman of childbearing potential
* Written informed consent after meeting with a study physician and ability and willingness to complete follow up.

Exclusion Criteria:

* No matching plasma donor (exact matching in both the ABO system and the Rh system is required)
* Unavailability of plasma
* Significant growth of alternative lower airway pathogen such as Streptococcus pneumoniae or Haemophilus influenzae in sputum
* Disease duration >8 Days
* Estimated glomerular filtration rate <60 (kidney failure stage III or more)
* Pregnancy (urinary-hcg), breast feeding,
* History of severe allergic reactions
* Inability to give informed consent
* Significantly compromised immunity.*

  * Compromised immunity includes but is not limited to treatment with major immunosuppressive agents including high dose corticosteroids, anti-tumor necrosis factor (TNF) agents, calcineurin inhibitors, mTOR inhibitors, lymphocyte depleting biological agents, chemotherapeutic anti neoplastic agents. Also patients with advanced HIV/AIDS, severe immunodeficiency such as hypoglobulinemia, decompensated liver cirrhosis and bone marrow transplant the last year will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Disease progression | 28 days
  Decrease in progression to requiring non-invasive or invasive ventilation

SECONDARY OUTCOMES:
Adverse events (AE) | The reporting period for AEs starts at inclusion and ends at the final follow-up visit 2 months after inclusion.
  Adverse reactions and serious adverse reactions. The safety of the intervention will be assessed with regard to AEs, baseline medical conditions, and findings from the physical examination and laboratory tests. Possible adverse events will be elicited using a modification and Swedish translation (appendix 6) of Common Terminology Criteria for Adverse Events v5.0 and they will be continuously reported to the sponsor. Adverse events related to convalescent plasma therapy shall be followed to assess reversibility.
Time ro resolution of fever and symptoms | Until discharged from the hospital, up to 2 months
  Measured daily until discharged from the hospital.
Clearance of viraemia | Evaluated daily until discharge, at day 28, and last measurement taken at 6 months of follow-up after inclusion.
  SARS-CoV-2 RNA detection by polymerase chain reaction (PCR) in blood or serum. Blood samples for immunological analyses and serology will be taken daily until discharge, on day 28, and at 6 months.
Inflammatory parameter C-reactive protein (CRP) | Until discharged from the hospital, up to 2 months
  Time to normalization of inflammatory parameter C-reactive protein (CRP). Blood sample for this marker will be taken daily until normalized or discharged from hospital.
Inflammatory parameter white blood cell count | Until discharged from the hospital, up to 2 months
  Time to normalization of inflammatory parameter white blood cell count (WBC). Blood sample for this marker will be taken daily until normalized or discharged from hospital.
Inflammatory parameter haemoglobin (Hb) | Until discharged from the hospital, up to 2 months
  Time to normalization of inflammatory parameter haemoglobin (Hb). Blood sample for this marker will be taken daily until normalized or discharged from hospital.
Inflammatory parameter Pro-calcitonin | Until discharged from the hospital, up to 2 months
  Time to normalization of inflammatory parameter Pro-calcitonin. Blood sample for this marker will be taken daily until normalized or discharged from hospital.
Inflammatory parameter Creatine Kinase | Until discharged from the hospital, up to 2 months
  Time to normalization of inflammatory parameter Creatine Kinase. Blood sample for this marker will be taken daily until normalized or discharged from hospital.
Antibody response to SARS-CoV-2 | Evaluated daily until discharge, at day 28, and last measurement taken at 6 months of follow-up after inclusion.
  Change in the antibody response to SARS-CoV-2 as measured in serum. Blood samples for immunological analyses and serology will be taken daily until discharge, on day 28, and at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Ursing, MD, PhD, Principal Investigator — Danderyd Hospital
Locations (1):
- Danderyd Hospital, Danderyd, Sweden

IPD SHARING:
Plan to Share IPD: Yes
We will be sharing data but data the management plan is being designed.